CLINICAL TRIAL: NCT01307358
Title: A Randomized Parallel Study Comparing the Interproximal Plaque and Gingivitis Effects of Three Interdental Cleaning Modalities
Brief Title: A Study Comparing the Interproximal Plaque and Gingivitis Effects of Three Interdental Cleaning Modalities
Acronym: PAU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Philips Oral Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DRC-0742
Record Dates: First submitted 2011-02-28; First posted 2011-03-02 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2017-01

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Manual Toothbrush + Sonicare Interproximal Cleaning Prototype (Experimental): Manual Toothbrush + Sonicare Interproximal (IP) Cleaning Prototype
  Interventions: Other: Sonicare Interproximal (IP) Cleaning Prototype
- Manual Toothbrush (Active Comparator): Manual Toothbrush
  Interventions: Other: Sonicare Interproximal (IP) Cleaning Prototype
- Manual Toothbrush + Floss (Active Comparator): Manual Toothbrush + Floss
  Interventions: Other: Sonicare Interproximal (IP) Cleaning Prototype
- Manual Toothbrush + Waterpik Ultra Water Flosser (Active Comparator): Manual Toothbrush + Waterpik Ultra Water Flosser
  Interventions: Other: Sonicare Interproximal (IP) Cleaning Prototype

INTERVENTIONS:
Other: Sonicare Interproximal (IP) Cleaning Prototype — Sonicare Interproximal (IP) Cleaning Prototype used to clean between the teeth 1 time a day in combination with brushing.

SUMMARY:
The purpose of this research study is to compare the interproximal plaque removal ability of Philips Sonicare Interproximal Cleaning Device to floss (Crest Glide) and Waterpik Waterflosser. In addition, we seek to learn more about the results of using this device on plaque accumulation and what biological processes influence the makeup of plaque and reduction of gingivitis.

DETAILED DESCRIPTION:
Primary Endpoint The primary endpoint of this study is the residual protein concentration in posterior sites following single use treatment with either manual toothbrush, manual toothbrush + Sonicare IP cleaning prototype, manual toothbrush + Waterpik Ultra Water Flosser or manual toothbrush + floss.

Secondary Endpoints Gingival bleeding index and Modified gingival index following single use treatment with either MTB, MTB + IP cleaning prototype, MTB + Waterpik Waterflosser or MTB + floss.

Comparisons of the concentration levels of 272 different pathogens between treatment groups

Biomarker profiles following the different treatment modalities

Safety endpoints based on adverse events and intraoral exam (soft tissue evaluation).

IP cleaning satisfaction questionnaire following treatment with either MTB, MTB + IP cleaning prototype, MTB + Waterpik Waterflosser or MTB + floss.

Expected Duration of Study The planned duration of a subject's participation in this study is approximately 2 weeks.

Discontinuation Criteria/Stopping Rules If in the opinion of the investigator, the health or safety of a subject is affected adversely by participation in the study or non-compliance to at-home oral hygiene regimen adversely effects test product familiarization or plaque regrowth, the subject will be removed.

Controls to Minimize Bias All eligible subjects will be randomized at Visit 1. Randomization of Subjects and Balance of Test Groups Subjects will be randomized to one of the four treatment groups according to a 1:1:1:1 ratio. Randomization will be stratified by gender to complete with approximately 68 subjects.

Blinding The examiner and laboratory personnel will be blinded.

Maintenance of randomization Codes In order to minimize bias, this study will be randomized and single blind - the Examiners performing the interproximal plaque sampling and gingivitis assessment are the designated blinded personnel. Unblinding of study data will not occur until after all study procedures have been completed.

Experimental Regimen and Product Labeling The devices used in this study are subject only to Class I (general controls) and considered exempt from the premarket notification procedures and not subject to section 510(k), 515, or 520(m,) of the FDC Act in order to be legally marketed. Thus, the study does not meet the definition of an Applicable Clinical Trial.

Each subject will receive an ADA Reference manual toothbrush, timer, dentifrice and, if assigned, an IP cleaning device (either Sonicare Prototype, Crest Glide Floss or Waterpik Ultra Water Flosser (WP 100) with the Classic Jet Tip). Subjects are to brush twice daily for two minutes and, if assigned, use their IP cleaning device once daily, in the evening, after toothbrushing. The Directions for Use for all devices can be found in the protocol Appendices and should be reviewed with the subjects who shall demonstrate proper usage at the time of product assignment.

Methods and Treatments not Permitted on Study Once enrolled on-study, the use of any additional oral hygiene treatments and aids other than those prescribed is prohibited. A list of prohibited devices and aids includes but is not limited to mouthwash, chewing gum, whitening products, non-assigned interproximal cleaning aids/devices or breath films. The use of any dentifrice other than that dispensed at Visit 2 is prohibited. In the event that an enrolled subject requires dental care outside the scope of the study, he/she will be discontinued from the trial.

The use of antibiotics or antibacterial agents while participating on the study is also prohibited and subjects who are required to use them will be removed from the dataset for endpoint analysis. The use of prescription strength and repeat dose of non-steroidal anti-inflammatories and anticoagulants (including Aspirin) for longer than 2 days is also prohibited.

All deviations from the prescribed treatment will be documented and continued eligibility will be reassessed.

Determination of Sample Size Sample size justification is based on considerations of statistical power for detecting a difference in mean residual protein concentration (RPC) between the manual toothbrush group and the manual toothbrush + Sonicare Interproximal (IP) Cleaning Prototype group. A sample size of 17 per group at visit 3 (the anticipated sample size after allowance for dropout) will provide 80% power for detecting a difference in mean RPC between groups of 4.71 (µg/ml) assuming a subject-level standard error of the average of two RPC measurements of 4.76 (the square of this standard error is the variance determined from assuming an RPC IP site-specific standard deviation of 6.15, and an intramouth correlation of the two RPC measurements of 0.2, as estimated from a statistical model (see 8.6) for preliminary data that adjusts for baseline RPC).

ELIGIBILITY:
Inclusion Criteria:

* are in good/excellent health
* are 18 - 70 years old
* have abstained from all oral care in the 12 hours prior to their scheduled appointment, but no more than 18 hours prior
* have abstained from consumption of apples and other sticky fruits in the 12 hours prior to their appointment
* have a minimum of 20 natural teeth (excluding 3rd molars)
* have 2 qualifying Interproximal Unit test sites in each posterior quadrant from 3 approximating teeth : The following are the IU test site qualifiers:
* Each IU test site shall consist of two adjacent teeth with un-restored interproximal surfaces with a closed contact. (Note: restorations are permissible if they do not interfere with plaque and GCF sampling as determined by examiner discretion)
* IU test sites of choice are as follows in the order of preference:
* Molar/premolar
* Premolar/premolar
* Molar/molar
* molar/canine
* have PPD ≤ 4mm at all four sites within each interproximal unit test site
* have ≥ 20 bleeding sites (whole mouth) as determined by the Gingival Bleeding Index
* have provided written informed consent and are willing to participate and be available at all times required for participation
* are willing and able to fully understand and comply with the written and verbal study instructions provided in English
* agree to return all study materials at the final visit

Exclusion Criteria:

* have systemic diseases, Down's syndrome, or known AIDS/HIV;
* Have Diabetes
* are a smoker
* are pregnant or nursing by subject report;
* have a cardiac pacemaker or AICD
* are undergoing or require extensive dental or orthodontic treatment;
* have had oral or gum surgery in the previous 2 months;
* require antibiotic treatment for dental appointments;
* have used antibiotics within 4 weeks of enrollment
* are currently using prescription-dose anti-inflammatory medications or anticoagulants (including aspirin)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
residual protein concentration in posterior sites | 2 weeks

SECONDARY OUTCOMES:
GBI and MGI | 2 weeks
  GBI and MGI following single use treatment with either MTB, MTB + IP cleaning prototype, MTB + Waterpik Waterflosser or MTB + floss.
  Comparisons of the concentration levels of 272 different pathogens between treatment groups Biomarker profiles following the different treatment modalities Safety endpoints based on adverse events and intraoral exam (soft tissue evaluation).
  IP cleaning satisfaction questionnaire following treatment with either MTB, MTB + IP cleaning prototype, MTB + Waterpik Waterflosser or MTB + floss.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Offenbacher, DDS,PhD,MMS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- GO Health Center, University of North Carolina, Chapel Hill, North Carolina, United States